CLINICAL TRIAL: NCT02358616
Title: An Exploratory Study of Potential Sources of Efficacy Dilution in the VOICE Trial
Brief Title: An Exploratory Study of Potential Sources of Efficacy Dilution in the VOICE Trial (MTN-003)
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-003D; 5UM1AI068633 (NIH); 11893 (Other Grant/Funding Number: DAIDS Protocol ID)
Record Dates: First submitted 2013-09-05; First posted 2015-02-09 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: HIV Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Former VOICE (MTN-003) participants: Qualitative interviews and focus group discussions conducted on former VOICE participants. All participants to receive interviews.

SUMMARY:
This study is primarily exploratory and is designed to both identify factors that may have affected participant adherence to study product in VOICE, and describe how sexual behaviors, such as anal sex, may have had an effect on product efficacy. As such there is no specific hypothesis that is being tested.

DETAILED DESCRIPTION:
MTN-003D will use qualitative in-depth interviews and/or focus group discussions with VOICE participants to explore study product adherence and/or anal sex behaviors in greater depth than was measured quantitatively during trial participation. The study approach is designed to encourage honesty and to minimize socially desirable responses, which may have affected participants' ability/willingness to accurately report during the trial. An in-depth and candid understanding of the various behavioral factors that contribute to the dilution of efficacy may assist in the interpretation of VOICE trial results and inform future studies.

In light of VOICE's divergent results, MTN-003D will explore the potential factors that may have contributed to efficacy dilution in the trial. MTN-003D, was initially designed after the early closure of the oral and vaginal tenofovir arms, and sought to explore those factors contributing to the dilution of efficacy using qualitative methods (Stage 1). Given the subsequent release of VOICE results in February of 2013 and the availability of drug PK data, Stage 2 of MTN-003D has been designed to explore factors influencing adherence in greater depth, including HIV risk perception and motivation to join the trial.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to perform the study procedures
* Able and willing to provide informed consent in one of the MTN-003D study languages
* Participated in VOICE and received at least three consecutive months of study product at any time during VOICE trial participation
* Stage 2 participants must have pharmacokinetic data available Note: Women from Stage 1 who have PK data available will be considered eligible for Stage 2

Exclusion Criteria:

* Has any condition that, in the opinion of the Investigator or Record(IoR)/ designee:

  * would preclude informed consent
  * make study participation unsafe
  * complicate interpretation of study outcome data
  * otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Former VOICE (MTN-003) participants
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Contextual issues affecting product use | End of Study
  To explore larger contextual issues and specific aspects of the VOICE trial that positively and negatively affected participants' actual and reported product use.

SECONDARY OUTCOMES:
Explore risk perceptions and motivation to join VOICE study | End of Study
  To explore participants' risk perceptions and motivations to participate in VOICE and the association of these factors with product use or non-use in a prevention trial setting.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane van der Straten, PhD, Study Chair — RTI International
Locations (5):
- South Africa (2):
  - Isipingo Clinical Research Site, Durban, KwaZulu-Natal
  - Overport Clinical Research Site, Durban, KwaZulu-Natal
- Makerere University - Johns Hopkins University Research Collaboration Clinical Research Site, Kampala, Uganda
- Zimbabwe (2):
  - Seke South Clinical Research Site, Harare
  - Zengeza 3 Clinical Research Site, Harare

REFERENCES:
- [Result] Simoni JM, Beima-Sofie K, Amico KR, Hosek SG, Johnson MO, Mensch BS. Debrief Reports to Expedite the Impact of Qualitative Research: Do They Accurately Capture Data from In-depth Interviews? AIDS Behav. 2019 Aug;23(8):2185-2189. doi: 10.1007/s10461-018-02387-3. PMID 30666522
- [Result] van der Straten A, Montgomery ET, Musara P, Etima J, Naidoo S, Laborde N, Hartmann M, Levy L, Bennie T, Cheng H, Piper J, Grossman CI, Marrazzo J, Mensch B; Microbicide Trials Network-003D Study Team. Disclosure of pharmacokinetic drug results to understand nonadherence. AIDS. 2015 Oct 23;29(16):2161-71. doi: 10.1097/QAD.0000000000000801. PMID 26544581
- [Derived] Katz AWK, Mensch BS, Woeber K, Musara P, Etima J, van der Straten A. Understanding women's motivations to participate in MTN-003/VOICE, a phase 2b HIV prevention trial with low adherence. BMC Womens Health. 2019 Jan 25;19(1):18. doi: 10.1186/s12905-019-0713-6. PMID 30683103
- [Derived] Luecke EH, Cheng H, Woeber K, Nakyanzi T, Mudekunye-Mahaka IC, van der Straten A; MTN-003D Study Team. Stated product formulation preferences for HIV pre-exposure prophylaxis among women in the VOICE-D (MTN-003D) study. J Int AIDS Soc. 2016 May 30;19(1):20875. doi: 10.7448/IAS.19.1.20875. eCollection 2016. PMID 27247202